CLINICAL TRIAL: NCT05983913
Title: Effects of Cognitive-motor Training Using a Wearable Sensor-based Interactive System on Cognitive and Motor Performance in Older Adults.
Brief Title: Effects of Wearable Sensor-based Interactive Cognitive-motor Training in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Jihye Jung, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2023-06-020-001
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Decline, Mild; Cognition Disorders in Old Age; Subjective Memory Decline
Keywords: cognitive-motor training; cogntion; physical function; older adults; interactive system; wearable sensor
MeSH Terms: conditions — Cognitive Dysfunction; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-group randomized study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive-motor training group (Experimental): Participants will receive 50 minutes of cognitive-motor training twice per week for 6 weeks. The cognitive-motor training program uses a wearable sensor-based interactive system to perform cognitive tasks in a large space without the constraints of physical movement. Participants wear a wearable sensor-based device on their dominant arm or leg and use an interactive system to perform cognitive-motor tasks.
  Interventions: Behavioral: cognitive-motor training
- cognition training group (Experimental): Participants will receive 50 minutes of cognitive training twice a week for 6 weeks. The cognitive training program will be delivered in booklet form, and participants will perform the cognitive tasks of the cognitive-motor training in a seated position with no physical movement.
  Interventions: Behavioral: cognition training

INTERVENTIONS:
Behavioral: cognitive-motor training — The cognitive-motor training program consists of five cognitive tasks related to concentration, reaction time, and executive function, combined with physical exercises using an interactive system. The five tasks include: (1) number sequence, (2) number-word sequence, (3) card matching games, (4) memorizing numbers, and (5) route-finding games.
  Arms: cognitive-motor training group
Behavioral: cognition training — The intervention consists of five cognitive tasks (memory, attention, spatial and temporal perception) with difficulty levels adapted to the individual's cognitive abilities.
  Arms: cognition training group

SUMMARY:
* Based on research showing that cognitive-motor training programs help improve cognition in older adults with mild cognitive impairment, this program uses an interactive system to combine cognitive training with exercise.
* The interactive system consists of wearable sensors and has the advantage of cognitive training without space constraints, and the cognitive training program consists of a total of five developed cognitive training games.
* The program is expected to improve the cognitive abilities of the elderly and improve their physical abilities.

DETAILED DESCRIPTION:
The proposed study will conduct a randomized controlled trial to compare the effects of a cognitive-motor training program using a wearable sensor-based interactive system on the cognitive and physical abilities of older adults in the community. Study participants will be randomly assigned to receive one of two interventions: (a) motor-cognitive training (b) cognitive training. All interventions will last 50 minutes and will be delivered twice a week for 6 weeks. To determine the effectiveness of the interventions, the primary outcome will assess PFC activity and cognition, and the secondary outcome will assess aerobic capacity, balance, upper extremity muscle strength, lower extremity muscle strength, and instrumental activities of daily living tasks. All assessments will be administered one week before and one week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling seniors age 65 and older
* MMSE-K 18 or less

Exclusion Criteria:

* People of Hospitalized or institutionalized
* People diagnosed with Alzheimer's disease
* People diagnosed with vascular dementia
* People with musculoskeletal conditions that make physical activity difficult
* People with dizziness that makes physical activity difficult
* People with a wound or bleeding in the head

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Change in prefrontal cortex activation | change from baseline to 6 week post intervention
  Activation of the prefrontal cortex will be assessed by changes in HbO, and differences in PFC activity will be identified during cognitive tasks (memory, attention, and visuospatial cognition) before and after the assessment.
Change in cognition | change from baseline to 6 week post intervention
  For cognitive assessment, we will use the Montreal Cognitive Assessment (MoCA). The MoCA is a cognitive assessment tool used to identify MCI that assesses multiple cognitive domains, including memory, attention, language, visuospatial skills, executive function, and orientation to time and place.

SECONDARY OUTCOMES:
Change in Aerobic capacity | change from baseline to 6 week post intervention
  Aerobic capacity is measured using the 6-minute walk test (6MWT). The 6MWT measures the distance a subject can walk in six minutes. You can take as many breaks as you like and the examiner can provide a chair. The examiner records the distance you walk in six minutes, the number of breaks you take, and the duration of the breaks.
Change in dynamic balance function 1 | change from baseline to 6 week post intervention
  The Four Square Step Test (FSST) is used to assess dynamic balance ability. The FSST consists of stepping safely and as quickly as possible, without touching the sticks, over four sticks placed in a criss-cross configuration on the floor, and is scored by recording the time in seconds.
Change in dynamic balance function 2 | change from baseline to 6 week post intervention
  Dynamic balance is assessed using the Functional Reach Test (FRT). The FRT measures the distance (in centimeters) that the head of the third metacarpal of the hand moves by extending the arm forward without moving the foot from a standing position.
Change in static balance function | change from baseline to 6 week post intervention
  To assess static balance, using the Single Leg Stance Test (SLS). The SLS measures the number of seconds standing on one leg with hands on hips and eyes open.
Change in upper extremity strengthen | change from baseline to 6 week post intervention
  Upper extremity strength is assessed with the arm curl test. On women perform a biceps curl with a 2.3 kg dumbbell and men with a 3.6 kg dumbbell. They are seated in a chair with no armrests or backrest. Scoring is based on the number of repetitions performed in 30 seconds.
Change in grip strengthen | change from baseline to 6 week post intervention
  Grip strength is measured using a dynamometer and the subject is seated in a chair with arms extended, natural rotation, elbow flexed 90 degrees, forearm at natural angle and wrist in dorsiflexion between 0 and 30 degrees. The subject is then asked to grip the dynamometer for 3 seconds and the average value (kg) over 3 trials is recorded.
Change in lower extremity strengthen | change from baseline to 6 week post intervention
  Lower extremity strength is assessed using the 5 sit to stand test (5xSST). The 5xSST measures the number of seconds a subject can go from sitting to standing and back to sitting five times, with the shorter the time, the better the strength.
Change in Instrumental Activity of Daily Living(IADLs) | change from baseline to 6 week post intervention
  IADLs require higher cognitive skills than basic activities of daily living, and IADLs can detect functional changes in the early stages of dementia. Instrumental IADLs are assessed using the Functional Activities Questionnaire (FAQ). The FAQ can differentiate between Mild cognitive impairment(MCI) and mild Alzheimer's disease(AD).

CONTACTS AND LOCATIONS:
Locations (1):
- Mapo senior welfare center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No